CLINICAL TRIAL: NCT03722875
Title: A Single Arm Pilot Study of Programmed Cell Death Drotein 1 Antibody (PD-1） SHR-1210 Combined With Apatinib Mesylate in Patients With Intermediate And Advanced-Stage Hepatocellular Carcinoma After Radical Hepatectomy
Brief Title: SHR-1210 Plus Apatinib in Patients With Hepatocellular Carcinoma After Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSGY-PA-1809
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab; spartalizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210+ apatinib (Experimental): SHR-1210 (200mg fixed dose every 3 weeks, one cycle is three weeks, total
  1 year ) will be administered as an intravenous infusion over 30 minutes.
  apatinib 250 mg qd ， one cycle is three weeks, total 1 year
  Interventions: Drug: SHR-1210; Drug: apatinib

INTERVENTIONS:
Drug: SHR-1210 — SHR-1210 is a humanized anti-PD1 IgG4 monoclonal antibody.
  Other Names: Anti-PD-1 Antibody
Drug: apatinib — Apatinib is a selective VEGFR2 inhibitor

SUMMARY:
SHR-1210 is a humanized anti-PD1 Immunoglobulin G4 (IgG4) monoclonal antibody. This is an open- label，single center ，non-randomized ，Single Arm Exploratory Study . This clinical study is an investigator-initiatedclini-cal trial（IIT ）.The objective of this study is to evaluate the efficacy and safety of adjuvant therapy with anti-PD-1 antibody SHR-1210 and apatinib in patients with Barcelona Clinic Liver Cancer (BCLC) B&C stage hepatocellular carcinoma after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. age:18-75 years, male or femal.
2. Hepatocellular carcinoma confirmed by histopathology, Child-Pugh A .
3. BCLC staging is stage B or C, preoperative assessment of no extrahepatic metastases.
4. ECOG Performance Status 0-1.
5. Alpha-fetoprotein (AFP) decreased to normal，3-4 weeks after surgery. If it is not normal, it must be checked that there is no clear lesion in MRI or CT.
6. Adequate organ function.
7. Patient has given written informed consent.

Exclusion Criteria:

1. No anti-tumor treatment for hepatocellular carcinoma, including chemotherapy and topical treatment, before surgery.
2. Known history of hypersensitivity to macromolecular protein preparation or any components of the SHR- 1210 formulation.
3. Tumors are not completely removed, or postoperative pathology suggests non-hepatocellular carcinoma or other malignant components;
4. Subjects with any active autoimmune disease or history of autoimmune disease
5. Uncontrolled clinically significant heart disease, including but not limited to the following: (1) > NYHA II congestive heart failure; (2) unstable angina, (3) myocardial infarction within the past 1 year; (4) clinically significant supraventricular arrhythmia or ventricular arrhythmia requirement for treatment or intervention;
6. Active infection or an unexplained fever > 38.5°C during screening or before the first scheduled day of dosing (subjects with tumor fever may be enrolled at the discretion of the investigator);
7. Received a live vaccine within 4 weeks of the first dose of study medication.
8. Pregnancy or breast feeding.
9. Decision of unsuitableness by principal investigator or physician-in- charge.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
relapse-free survival(RFS) | 1 year
  from the date of enrollment to tumor recurrence or Death
Overall survival(OS) | 3 years
  the date of Death of any causes since the date of enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided